CLINICAL TRIAL: NCT06004323
Title: Digital Health Literacy on COVID-19 for All: Co-creation and Evaluation of Interventions for Ethnic Minorities and Chinese People With Chronic Illnesses in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Angela Leung, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSEARS20210902004
Record Dates: First submitted 2023-08-21; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Digital Health Literacy; COVID-19
Keywords: Digital health literacy; COVID-19; Ethnic minorities; Chinese people with chronic illnesses
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a single-blinded, randomized controlled trial that outcome assessors will be prevented from having knowledge of the interventions assigned to individual participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital health literacy intervention (Experimental): The interventions will be developed based on the Best Practices for Digital Health Literacy, WHO health literacy toolkits and the findings of the interviews. The content to be covered in the intervention will include news about vaccines; alerts about COVID-19 preventive measures; guidelines on social distancing, COVID-19 screening test arrangements, vaccination and compulsory quarantines; COVID-19-related law enforcement; and self-monitoring of COVID-19 symptoms
  Interventions: Behavioral: Digital health literacy intervention
- Control (No Intervention): No intervention will be provided to the control group

INTERVENTIONS:
Behavioral: Digital health literacy intervention — Participants from the intervention group will be invited to join virtual or face-to-face training, watch short videos on social media, participate in virtual bi-weekly group discussion, and fill in questionnaires for five times during the course of the study
  Arms: Digital health literacy intervention

SUMMARY:
During the pandemic, people are anxious for information, and electronic platform serves the purpose of having first-hand health information and spreading it to massive population within a short time. However, the source and credibility of the influx of online information are hard to be verified. Digital health literacy (DHL) is the capacity to access, understand, evaluate, and apply health information from electronic sources, which is an important attribute that everyone should possess. Recent studies from our group in Hong Kong have shown that, during the COVID-19 pandemic, DHL is an issue facing people of all ages, especially ethnic minorities (EMs), people with chronic illnesses (PWCI), and professional and lay caregivers (CGs). Considering that, the present research project aims to co-create DHL interventions with these three groups of people to meet their specific needs in DHL, in addition, to assess the efficacy of the DHL interventions on eHealth literacy, vaccine literacy, and actions taken for COVID-19 prevention. The present research is a 4-year project, involving three phases. Phase 1 involves focus group interviews and cognitive interviews with the three groups of people for developing interventions and evaluating the proposed interventions. Phase 2 involves individual interviews with the three groups of people for testing the feasibility and acceptability of the interventions. Phase 3 involves a 6-month longitudinal quantitative research, testing for the efficacy of the interventions in three dimensions: literacy, attitude, and behavior. Participants from the three groups will be invited to join virtual or face-to-face training, watch short videos on social media, participate in virtual bi-weekly group discussion, and fill in questionnaires for five times during the course of the study. This co-creation of new knowledge by stakeholders and researchers is expected to increase the uptake of the research outcomes and adoption of the DHL interventions.

ELIGIBILITY:
Inclusion Criteria:

* ethnic minorities (EMs), people with chronic illnesses (PWCI), and caregivers (CGs)
* able to use a computer, smartphone, or laptop to access the Internet at home

Exclusion Criteria:

* diagnosis of an acute psychotic disease or life-limiting condition; having a visual, auditory, or fine motor disorder.

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
eHealth Literacy Efficacy | baseline, 8-week post intervention, 4-week post follow-up, 8-week follow up, and 12 week follow up
  Measured by the eHealth Literacy scale (eHEAL), an 8-item self-reported efficacy scale scored on a 5-point Likert scale

SECONDARY OUTCOMES:
Digital Health Literacy | baseline, 8-week post intervention, 4-week post follow-up, 8-week follow up, and 12 week follow up
  Measured by Digital Health Literacy Instrument
Vaccine literacy | baseline, 8-week post intervention, 4-week post follow-up, 8-week follow up, and 12 week follow up
  knowledge about and intention to receive the COVID-19 vaccine
Knowledge, attitudes, and practices towards COVID-19 | baseline, 8-week post intervention, 4-week post follow-up, 8-week follow up, and 12 week follow up
  Assess knowledge, attitudes, and practices towards COVID-19

IPD SHARING:
Plan to Share IPD: No
Data can be obtained from principal investigator.